CLINICAL TRIAL: NCT03055520
Title: Arithmetic Calculation Training With the Kumon Errorless Learning Method for Cognitive Rehabilitation of Patients With Schizophrenia: a Randomized Controlled Trial
Brief Title: Arithmetic Training With the Kumon Method for Cognition in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mario R. Louza, MD, PhD, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cognition schizophrenia
Record Dates: First submitted 2017-02-10; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognition; arithmetic training; Kumon method
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arithmetic training (Kumon method) (Experimental)
  Interventions: Other: cognitive training
- nonspecific recreation (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Other: cognitive training — The Kumon method (www.kumon.com) of arithmetic calculation employs the errorless-learning (EL) strategy and consists of a structured, hierarchical series of exercises, beginning with simple ones (e.g. addition and subtraction) and then proceeding to more complex exercises (e.g. advanced algebra, calculus).
  Arms: arithmetic training (Kumon method)
Other: placebo — nonspecific recreation including befriending and free simple activities.
  Arms: nonspecific recreation

SUMMARY:
A randomized placebo-controlled trial of arithmetic training (with the Kumon Method) as an errorless learning method for improvement of cognition in schizophrenia. Outpatients were included after signing an informed consent. The trial consisted of 48 sessions of arithmetic training (twice a week, for 6 months) or placebo (nonspecific recreation, 48 sessions). The patients were evaluated with a neuropsychological battery at baseline, after 6 months (end of intervention) and after 12 months after baseline. The Positive and Negative Syndrome Scale (PANSS) and the Personal and Social Performance scale (PSP) were applied at baseline, after 6 months (end of intervention) and 12 months after baseline. Primary outcome was the performance on three cognitive domains (attention, executive functions and working memory).

ELIGIBILITY:
Inclusion Criteria:

* Literate (≥5 years of formal education).
* Diagnostic criteria for schizophrenia according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-IV-TR).
* Clinically stable, with constant antipsychotic medication regimen for ≥8 weeks before screening
* No hospitalizations in the last 6 months.

Exclusion Criteria:

* Other Axis I psychiatric disorders, substance abuse or dependence.
* History of head trauma or other neurologic diseases.
* Severe or uncontrolled medical diseases, history of mental retardation or attendance in special-education classes,
* Suicide risk
* Participation in any other kind of psychosocial intervention.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
improvement in attention | change from baseline to 6 months and to 12 months
  neuropsychological battery
improvement in working memory | change from baseline to 6 months and to 12 months
  neuropsychological battery
improvement in executive function | change from baseline to 6 months and to 12 months
  neuropsychological battery

SECONDARY OUTCOMES:
psychopathology | change from baseline to 6 months and to 12 months
  Evaluation with the Positive and Negative Syndrome Scale (PANSS)
functioning | change from baseline to 6 months and to 12 months
  Evaluation with the Personal and Social Performance (PSP) scale

IPD SHARING:
Plan to Share IPD: Undecided